CLINICAL TRIAL: NCT07235137
Title: A Phase 1, Single Arm Study to Evaluate the Pharmacokinetics Following Single Dose of PF-07817883 (Ibuzatrelvir) in Healthy Chinese Adult Participants.
Brief Title: A Study to Learn How the Study Medicine Called Ibuzatrelvir is Taken up Into the Blood in Healthy Chinese Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: C5091002
Record Dates: First submitted 2025-11-14; First posted 2025-11-19 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Healthy Participant
Keywords: severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2); coronavirus disease 2019 (COVID-19)
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ibuzatrelvir (Experimental): Ibuzatrelvir will be given by mouth to adult Chinese healthy volunteers
  Interventions: Drug: Ibuzatrelvir

INTERVENTIONS:
Drug: Ibuzatrelvir — Ibuzatrelvir will be given by mouth to adult Chinese healthy volunteers
  Other Names: PF-07817883

SUMMARY:
A study to learn how the study medicine called Ibuzatrelvir is taken up into the blood in healthy Chinese adults.

DETAILED DESCRIPTION:
To evaluate the PK profile of ibuzatrelvir after administration in Chinese healthy participants

ELIGIBILITY:
Inclusion:

* Male and female participants aged from 18 years old or older at screening who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and ECG.
* BMI of 16-32 kg/m2 (both inclusive); and a total body weight >45 kg (99 lbs.).
* Chinese male and female participants are defined as individuals currently residing in mainland China who were born in China and have both parents of Chinese descent.

Exclusion:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Any condition possibly affecting drug absorption (e.g., gastrectomy, cholecystectomy).
* History of HIV infection, hepatitis B, or hepatitis C; positive testing for HIV, HBsAg, or HCVAb. Hepatitis B vaccination is allowed.
* Any medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality or other conditions that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
* Use of prescription or nonprescription drugs and dietary and herbal supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study intervention.
* Previous administration of an investigational product (drug or vaccine) within 30 days or 5 half-lives preceding the first dose of study intervention used in this study (whichever is longer). Participation in studies of other investigational products (drug or vaccine) at any time during participation in this study.
* A positive urine drug test. A single repeat for positive drug screen may be allowed.
* Pregnant or breastfeeding women.
* Screening supine BP ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic) for participants <60 years; and ≥150/90 mm/Hg for participants ≥60 years old, following at least 5 minutes of supine rest. If systolic BP is ≥140 or 150 mm Hg (based on age) or diastolic ≥90 mm Hg, the BP should be repeated 2 more times, and the average of the 3 BP values should be used to determine the participant's eligibility.
* Standard 12-lead ECG that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results (e.g., QTcF >450 ms, complete LBBB, signs of an acute or indeterminate- age myocardial infarction, ST segment and/or T wave changes suggestive of myocardial ischemia, second- or third- degree AV block, or serious bradyarrhythmia or tachyarrhythmias). If QTcF exceeds 450 ms, or QRS exceeds 120 ms, the ECG should be repeated twice and the average of the 3 QTcF or QRS values used to determine the participant's eligibility. Computer-interpreted ECGs with abnormal findings should be overread by a physician experienced in reading ECGs before excluding a participant.
* Participants with ANY of the following abnormalities in clinical laboratory tests at screening, as assessed by the study-specific laboratory and confirmed by a single repeat test, if deemed necessary: ALT, AST, Bilirubin ≥1.5× ULN

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2025-10-16 (Actual); Primary Completion 2025-11-21 (Actual); Study Completion 2025-11-21 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | up to Day 3
AUCinf | up to Day 3
Terminal phase half-life (t½) | up to Day 3

SECONDARY OUTCOMES:
Adverse events and severe adverse events | up to Day 3
Incidence of abnormal and clinically relevant changes in vital signs | up to Day 3
Incidence of abnormal and clinically relevant changes in electrocardiogram | Up to Day 3
Incidence of abnormal and clinically relevant changes in laboratory assessments | Up to Day 3

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C5091002